CLINICAL TRIAL: NCT07307339
Title: The Acute Effects of Blood Flow Restriction on Ankle Muscle Reaction Time and Proprioception in Healthy Individuals
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Melike Tugran, MD, Uludag University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-15/31
Record Dates: First submitted 2025-11-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Ankle Proprioception; Blood Flow Restriction
Keywords: ankle; proprioception; blood flow restriction
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Arm 1: Experimental - Blood Flow Restriction Participants perform balance and proprioception tests under lower-limb blood flow restriction at 60% arterial occlusion pressure.
  Arm 2: Sham Comparator - Sham Blood Flow Restriction Participants perform the same balance and proprioception tests with sham blood flow restriction at 20 mmHg.
  This is a randomized crossover study, and all participants complete both conditions in a randomized order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Flow Restriction (Experimental): Participants perform balance/proprioception tests under lower limb blood flow restriction at % 60 AOP.
  Interventions: Other: Blood Flow Restriction
- Sham BFR (Sham Comparator): Sham BFR Description: Participants perform the same tests with sham(20 mmHg) blood flow restriction
  Interventions: Other: Sham Blood Flow Restriction

INTERVENTIONS:
Other: Blood Flow Restriction — Arm Description: Participants perform balance/proprioception tests under lower limb blood flow restriction at % 60 AOP.
  Arms: Blood Flow Restriction
Other: Sham Blood Flow Restriction — Sham BFR Description: Participants perform the same tests with sham(20 mmHg) blood flow restriction
  Arms: Sham BFR

SUMMARY:
his randomized controlled crossover study aims to investigate the acute effects of lower limb blood flow restriction (BFR) on ankle joint proprioception, postural control, and muscle activation in healthy adults. Each participant will complete test sessions under BFR (60% individualized arterial occlusion pressure) and control (20 mmHg sham) conditions. Outcome measures include joint position sense, kinesthesia, static and dynamic balance performance, and electromyographic (EMG) activity and reaction times of selected lower limb tibialis anterior and peroneus longus muscles.

DETAILED DESCRIPTION:
Lateral ankle sprains are among the most common musculoskeletal injuries and may lead to chronic ankle instability (CAI), partly due to impaired proprioception and neuromuscular control. Blood flow restriction (BFR) training is widely used to augment muscular adaptations with low external loads; however, its acute effects on joint proprioception and sensorimotor control, particularly at the ankle joint, remain unclear and may be detrimental under certain conditions. This randomized controlled crossover trial will examine the effects of a single-session lower limb BFR application on ankle joint position sense, kinesthesia, static and dynamic balance, and EMG-based reaction time and activity of lower limb muscles in healthy adults. Participants aged 18-40 years without recent ankle sprain, neuromuscular, cardiovascular, or thromboembolic disease will undergo standardized proprioception tests using an isokinetic dynamometer, static balance tests on a force platform, Y-balance test, and inversion simulation platform assessments under BFR (60% arterial occlusion pressure) and low-pressure control (20 mmHg) conditions. Individual arterial occlusion pressure (AOP) will be determined using Doppler ultrasound, and BFR will be applied with a pneumatic cuff at the most proximal thigh. All measurements will be performed on the dominant lower limb with sessions scheduled at the same time of day to minimize circadian variability. The primary hypothesis is that acute lower limb BFR will worsen ankle joint proprioception and sensorimotor control compared with the control condition, potentially indicating a transient increase in injury risk during BFR-assisted activities.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40 years
* No known neuromuscular or cardiovascular disease

Exclusion Criteria:

* History or presence of cardiac, coronary artery, or peripheral arterial disease
* Presence or history of varicose veins, hypertension, diabetes mellitus, or pulmonary disease
* History of pulmonary embolism or deep vein thrombosis
* Use of medications affecting the central nervous or cardiovascular systems
* Use of oral contraceptives or anticoagulants
* Pregnancy
* Open wounds or significant scar tissue at the cuff application site
* History of lower extremity musculoskeletal injury or surgery
* Any neurological, vascular, or systemic condition that may interfere with test performance

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Change in Ankle Joint Position Sense Error (degrees) | day 1 and day 2
  Absolute error (degrees) between target and reproduced angles during passive and active joint position sense tests in inversion and plantar flexion, measured with an isokinetic dynamometer.
Static Balance Performance | day 3
  Center of pressure path length (mm) in single-leg and tandem stance with eyes open/closed on force platform (HUR SmartBalance).
Change in Kinesthesia Threshold (degrees) | day 1 and day 2
  Minimal angular displacement (degrees) at which movement is first perceived in inversion and plantarflexion.
Static balance performance | day 3
  sway velocity (mm/s) in single-leg and tandem stance with eyes open/closed on force platform (HUR SmartBalance).
static balance performance | day 3
  sway area (mm^2) in single-leg and tandem stance with eyes open/closed on force platform (HUR SmartBalance).

SECONDARY OUTCOMES:
Y-Balance Test Reach Distances (cm) | day 4
  Anterior, posteromedial and posterolateral reach distances of the tested limb.
Peroneus Longus and Tibialis Anterior Reaction Time (ms) | day 4
  Time from onset of platform-induced inversion to EMG activation exceeding 2× resting activity.
Lower Limb EMG Activity (%MVIC) | day 4
  Mean EMG amplitude normalized to maximal voluntary isometric contraction values.

CONTACTS AND LOCATIONS:
Overall Officials: ufuk sekir, Study Director — Department of Sports Medicine, Bursa Uludağ University
Locations (1):
- Uludag University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No